CLINICAL TRIAL: NCT03751514
Title: A Human Controlled Infection Study to Establish a Safe, Reproducible and Practical Human Bordetella Pertussis Colonisation Model for the Identification of Correlates of Protection Against Colonisation (BPCCS)
Brief Title: Bordetella Pertussis Colonisation Challenge Study
Acronym: Periscope
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Southampton (Other)
Collaborators: Public Health England (Other Government); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RHM MED1396; 17/SC/0006 (Other: REC)
Record Dates: First submitted 2017-08-15; First posted 2018-11-23 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Whooping Cough
Keywords: Bordetella Pertussis
MeSH Terms: conditions — Whooping Cough | interventions — Azithromycin; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Human challenge study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase A - SI (Experimental): Phase A aims to determine a 'standard inoculum' dose (SI), which results in safe colonisation of 70% of volunteers.
  The SI will be identified in a dose escalating or de-escalating experiment commencing at 10-3 colony forming units B. pertussis administered intranasally. Each group of volunteers will be inoculated at half log-fold increasing/decreasing doses until the endpoint is reached. The experiment will be continued until the SI yields 10 subjects who are colonised at day 14.
  Intervention to be administered: Bordetella Pertussis B1917
  Interventions: Biological: Bordetella Pertussis B1917; Drug: Azithromycin 500 mg
- Phase B Inoculum (Experimental): Phase B, using study data from phase A, will be used to design a more practical model - if possible conducted partially in an outpatient setting, which will be conditional on safety and transmission evidence. The final protocol for phase B will be presented as a protocol amendment, it will be based on the SI and colonisation period identified in Phase A.
  The SI determined in phase A will be used for all volunteers and eradication therapy will be given after the colonisation period based on the data of phase A. Approximately 30 individuals will receive the intranasal SI and will be treated with azithromycin for three days at the end of the colonisation period.
  Intervention to be administered: Bordetella Pertussis B1917
  Interventions: Biological: Bordetella Pertussis B1917; Drug: Azithromycin 500 mg
- Phase B Sham (Experimental): Phase B, using study data from phase A, will be used to design a more practical model - if possible conducted partially in an outpatient setting, which will be conditional on safety and transmission evidence.
  Approximately 15 individuals will not receive the Bordetella Pertussis B1917, instead they will be given an intranasal sham of sterile saline and will be treated with azithromycin 500mg for three days at the end of the 'colonisation' period.
  Interventions: Drug: Azithromycin 500 mg; Other: Sterile Saline

INTERVENTIONS:
Biological: Bordetella Pertussis B1917 — The B. pertussis isolate to be used in this human colonisation model is strain B1917, which is representative of current isolates in Europe. The strain, isolated in 2000 from a Dutch patient with B. pertussis disease, expresses Prn, PT and Filamentous Haemagglutinin (FHA). This strain has been extensively characterised in the mouse model as well as by proteomics and transcriptomics and has a closed genome available. It is fully sensitive to azithromycin in vitro.
  Providing there are no safety concerns the standard inoculum (SI) will be identified in a dose escalating or de-escalating experiment commencing at 103 colony forming units administered intranasally.
  Other Names: Whooping cough bacteria
  Arms: Phase A - SI; Phase B Inoculum
Drug: Azithromycin 500 mg — To ameliorate risk of transmission of B. pertussis B1917 to the environment and household contacts, Azithromycin 500 mg once a day for 3 days will be given to eradicate colonisation with B. pertussis. The inoculum strain is fully sensitive to this antibiotic. Previous studies show that azithromycin eradicates colonisation in 97% of people in 48 hours.
  Other Names: Zithromax
Other: Sterile Saline — To compare against B. pertussis, some volunteers will be enrolled onto the Sham arm. These volunteers will not receive B. pertussis but instead be given sterile saline
  Other Names: Sham
  Arms: Phase B Sham

SUMMARY:
This is a prospective controlled human challenge study consisting of two phases; Phase A: Development of a B. pertussis human challenge model; pilot to establish the standard inoculum Phase B: Development of a modified B. pertussis human challenge model

DETAILED DESCRIPTION:
This study is part of work package 2 of the Periscope consortium. The Periscope consortium brings together internationally renowned scientists with many years of experience in B. pertussis research, clinical trials, bioinformatics, immunology and public health to promote scientific and technological innovation in pertussis vaccine development and to foster the creation of a laboratory and scientific network that facilitates the testing and helps expedite the development of novel pertussis vaccines in Europe. This study, the development of a human challenge model for B. pertussis, is one of the models that will accelerate the development and registration of novel pertussis vaccines and will provide samples for studies performed within the network.

This is a prospective controlled human challenge study consisting of two phases; Phase A: Development of a B. pertussis human challenge model; pilot to establish the standard inoculum The first aim of phase A is to determine a 'standard inoculum' (SI), which results in safe colonisation of 70% of volunteers. This level of colonisation of 70% has been selected so that baseline immune profiles of individuals who are, or are not colonised following challenge can be assessed and biomarkers of protection from colonisation identified. It is acknowledged that for the future use of the human challenge model for efficacy evaluation of experimental vaccine candidates, it would be optimal if the percentage of subjects successfully colonised were at least 70%. The SI will be identified in a dose escalating or de-escalating experiment commencing at 103 colony forming units B. pertussis administered intranasally. Each group of 5 volunteers will be sequentially inoculated at half log-fold increasing/decreasing doses until the endpoint is reached. The experiment will be continued until the SI yields 10 subjects who are colonised at day 14. Volunteers will be screened to exclude those with evidence of recent B. pertussis infection using anti-pertussis toxin (PT) immunoglobulin G (IgG) ELISA as evidence to allow evaluation of seroconversion. Following the challenge chemical, haematological and clinical parameters will be monitored and nasal swab samples will be cultured at regular intervals to assure safety of the volunteers and to identify the presence of B. pertussis. At day 14 after the challenge, or at the onset of symptoms, whichever occurs soonest, eradication therapy in the form of azithromycin 500 mg once a day for 3 days will be given. Further mucosal and blood samples will be taken over the follow up period of one year.

The second aim of phase A is to identify the 'colonisation period'; the earliest day after inoculation at which colonisation of the nasopharynx (as detected by culture) is observed in 100% of those volunteers who show seroconversion at day 28. This time period will be used to establish the length of participation required from volunteers in future studies. The colonisation period will be deemed biologically relevant if B. pertussis specific mucosal and systemic antibodies are elicited in people who are colonised for the colonisation period. A quantitative PCR assay to detect B. pertussis in nasopharyngeal samples will be evaluated to determine if this can provide more rapid information in addition to culture.

The third aim of phase A is to access environmental shedding of B. pertussis following nasal inoculation of healthy volunteers with B. pertussis. These shedding results will used to determine the length of admission and isolation in phase B. The shedding of B. pertussis by challenged volunteers will be assessed using personal aerosol samplers and environmental sampling. Efficacy of eradication therapy will be assessed.

Phase B: Development of a modified B. pertussis human challenge model In phase B the pilot study data from phase A will be used to design a more practical model, if possible conducted partially in an outpatient setting, which will be conditional on safety and transmission evidence. The final protocol for phase B will be presented as a protocol amendment, because it will be based on the standard inoculum and colonisation period identified in Phase A.

Volunteers in phase B will not be preselected to exclude those with evidence of recent B. pertussis infection. The standard inoculum determined in phase A will be used for all volunteers and eradication therapy will be given after the colonisation period based on the data of phase A. Approximately 30 individuals will receive the intranasal SI and as control group approximately 15 individuals will receive intranasal sham. Both groups will be treated with azithromycin for three days at the end of the colonisation period.

Aims:

* To confirm that the following parameters of the model in phase B are similar to that seen in phase A:

  * Volunteer safety
  * Colonisation rate
  * Colonisation period
  * Genetic/expression changes in B. pertussis during challenge
  * Environmental shedding
  * Efficacy of eradication therapy
* To compare the pattern of detection of B. pertussis in nasopharyngeal samples by qPCR to that seen in phase A.
* To assess B. pertussis-specific immunity before and after inoculating healthy volunteers with B. pertussis, comparing the data from successfully colonised participants with the data from those not colonised and the control group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of screening
* Fully conversant in the English language
* Able to communicate easily by both mobile telephone and text messaging
* Able and willing (in the investigator's opinion) to comply with all study requirements
* Written informed consent to participate in the trial
* Willingness to take a curative antibiotic regimen after inoculation with B. pertussis according to the study protocol
* Agreement to be admitted to the National Institute for Health Research (NIHR)-Clinical research facility (CRF) Southampton for 17 days for phase A (from inoculation until two days after the eradication therapy is given) and for the duration necessary for phase B, depending on phase A results
* Able to answer all questions on the informed consent quiz correctly

Exclusion Criteria:

* Individuals who have inviolable commitments within 3 months of discharge from the inpatient phase of the study to make contact with:

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
* Individuals who have household contacts working with

  1. unimmunised or partially immunised children and infants aged < 1 year
  2. pregnant women >32 weeks who have not received pertussis vaccination at least a week prior to contact
* Phase A only: Volunteers will be excluded from this study if they have evidence of recent exposure to B. pertussis, as determined by anti-PT IgG ELISA (>20 IU/mL)
* B. pertussis detected on nasopharyngeal swab taken before the challenge
* Individuals who have a signs of a current infection at the time of inoculation with B. pertussis
* Individuals who have participated in other interventional clinical trials in the last 12 weeks
* Individuals who have a history of receiving B. pertussis vaccination in the last 5 years
* Individuals who have a history of never being vaccinated against B. pertussis
* Current smokers defined as having had a cigarette/cigar in the last week.
* Use of systemic antibiotics within 30 days of or during the challenge
* Any confirmed or suspected immunosuppressive or immune-deficient state, including HIV infection; asplenia; recurrent, severe infections and chronic (more than 14 days) immunosuppressant medication within the past 6 months (topical steroids are allowed)
* Use of immunoglobulins or blood products within 3 months prior to enrolment
* History of allergic disease or reactions likely to be exacerbated by any component of the inoculum
* Contraindications to the use of azithromycin or macrolides
* Pregnancy, lactation or intention to become pregnant during the study
* Any clinically significant abnormal finding on biochemistry, haematology, toxicology or serological blood tests, urinalysis or clinical examination - in the event of abnormal test results, confirmatory repeat tests will be requested
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study or impair interpretation of the study data, for example recent surgery to the nasopharynx

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-05-22 (Actual); Primary Completion 2021-02-02 (Estimated); Study Completion 2021-02-02 (Estimated)

PRIMARY OUTCOMES:
Phase A - Inoculum Dose Determination | Up to volunteer visit Day 14
  The inoculum dose required to cause the safe colonisation of 70% of volunteers who are challenged. A starting inoculum of 10^3 bacteria will be used and incrementally increased until microbiologically proven Bp infection by positive culture of Bp from a nasopharyngeal swab (CFU/mL). Swabs are taken between time points day 0 and day 14 and compare with baseline.

SECONDARY OUTCOMES:
Phase A and B - Immune Responses to exposure to Bordetella pertussis | Up to volunteer visit Week 52
  Measure the antibody response (IU/L) of volunteers who receive the inoculum against the immune responses of those that receive the sham treatment.
Phase A - Accuracy of Inoculum Dosing Evaluation | Up to volunteer visit Day 7
  Measurement of the challenge dose (cfu/mL) actually given to volunteers by counting CFUs after culturing. This is done by culturing the remaining inoculum which has been given to the volunteers. Results are then compared with the prescribed dose (cfu/mL).
Phase A and B - Number of participants with Bp exposure-related adverse events as assessed by study specific adverse event grading system based on CTCAE v4.0 | Up to volunteer visit Day 365
  After inoculation with Bordetella pertussis, participants will be admitted in the research unit to monitor adverse events closely.
Phase A - Earliest Timepoint for Colonisation of the Nasopharynx | Up to volunteer visit Day 14
  The earliest day after inoculation at which colonisation of the nasopharynx (as detected by culture) is observed in 100% of those volunteers who subsequently seroconvert at day 28. Colonisation will be detected by positive culture of Bp from a nasopharyngeal swab taken between timepoints day 0 and 14
Phase A and B - Bacterial Dynamics after Challenge | Up to volunteer visit Day 14
  Microbiological assays to detect and characterise Bp after challenge in nasopharyngeal swabs (culture and qPCR), nasal wash (culture including semi-quantitative method using cfu count/mL, and precision quantification with qPCR)and sequencing of isolates
Phase A and B - Bacterial Dynamics after Challenge by culture | Up to volunteer visit Day 14
  Bp colonisation will be measured in nasopharyngeal swabs, nasal wash and throat swabs by culture using cfu count/mL
Phase A and B - Bacterial Dynamics after Challenge by PCR | Up to volunteer visit Day 14
  Bp colonisation will be measured in nasopharyngeal swabs, nasal wash and throat swabs by culture using cfu count/mL
Phase A - Environmental shedding of Bp | Day 0-16
  Air and mask samples will be collected of volunteers and cultured. Results will be expressed as cfu count
Phase A & B - Immune Response in nasal wash to Challenge | Up to volunteer visit Week 52
  Immunological laboratory assays to measure innate, humoral, cell-mediated and mucosal responses to challenge in nasal washes.
Phase A & B - Human Immune Response to Challenge in Saliva | Up to volunteer visit Week 52
  Antibody responses to challenge in saliva will be measured (Bp specific Immunoglobulin A (IgA) (IU/mL))
Phase A & B - Correlation of qPCR results with Culture Results after Challenge | Up to Day 16
  Comparison of qPCR results with culture results after challenge: Microbiological assays in nasopharyngeal swabs and nasal washes (culture, qPCR) taken between day 0 and 16

CONTACTS AND LOCATIONS:
Overall Officials: Robert C Read, MB MD FRCP, Principal Investigator — University of Southampton
Locations (1):
- NIHR Wellcome Trust Clinical Research Facility, Southampton General Hospital, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diks AM, de Graaf H, Teodosio C, Groenland RJ, de Mooij B, Ibrahim M, Hill AR, Read RC, van Dongen JJ, Berkowska MA; IMI-2 PERISCOPE Consortium. Distinct early cellular kinetics in participants protected against colonization upon Bordetella pertussis challenge. J Clin Invest. 2023 Mar 1;133(5):e163121. doi: 10.1172/JCI163121. PMID 36649086
- [Derived] de Graaf H, Ibrahim M, Hill AR, Gbesemete D, Vaughan AT, Gorringe A, Preston A, Buisman AM, Faust SN, Kester KE, Berbers GAM, Diavatopoulos DA, Read RC. Controlled Human Infection With Bordetella pertussis Induces Asymptomatic, Immunizing Colonization. Clin Infect Dis. 2020 Jul 11;71(2):403-411. doi: 10.1093/cid/ciz840. PMID 31562530